CLINICAL TRIAL: NCT04646213
Title: Managing Cancer and Living Meaningfully (CALM) in Primary Brain Tumor Patients
Brief Title: Managing Cancer and Living Meaningfully
Acronym: CALM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-20-16440; HM20020308 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Mood; Cancer Brain
MeSH Terms: conditions — Brain Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapy (Experimental): psychotherapeutic intervention
  Interventions: Behavioral: Managing Cancer and Living Meaningfully (CALM) Therapy

INTERVENTIONS:
Behavioral: Managing Cancer and Living Meaningfully (CALM) Therapy — 6 sessions of individualized CALM therapy

SUMMARY:
The purpose of this study is to pilot test an empirically supported psychotherapeutic intervention, Managing Cancer and Living Meaningfully (CALM). Researchers hope to better understand the potential benefits of this intervention on brain tumor patients' mood and quality of life. This may lead to improvements in doctor's understanding of how to enhance brain tumor patient's wellbeing and overall functioning.

DETAILED DESCRIPTION:
In this study, participants will be asked to do the following things:

1. Complete ~15-minute online surveys before the program, immediately after the program (4 months), and at follow-up (6 months). . Questions will ask about mood, anxiety, death distress, quality of social relationships, and satisfaction with life.
2. Meet with an interventionist six times (biweekly) for individual sessions via Zoom, lasting 50-60 minutes each. Sessions will be audio-recorded to ensure all participants receive the same information. Participants will be asked to only use first names.
3. Complete weekly ~5 minute online surveys after each session on satisfaction with the program.
4. Complete an exit interview by telephone approximately 1 month after the 6-session intervention. This exit interview will last approximately 15-30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* have a confirmed malignant brain cancer diagnosis via histopathology
* be a minimum of 2 weeks post-surgical resection or biopsy (if applicable)
* be primarily English speaking
* be age 18-89
* obtain >20 on the Telephone Interview for Cognitive Status (TICS)
* have current elevated depression or death anxiety symptoms
* have a reliable internet connection to participate in the Zoom therapy sessions

Exclusion Criteria:

* Major communication difficulties as determined by the research team which would prohibit psychotherapeutic interaction
* inability to meet with interventionist via an electronic device for telehealth intervention sessions
* inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2022-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashlee Loughan, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Individual level data will not be shared other researchers. Access to all data will be limited to study personnel.

REFERENCES:
- [Derived] Loughan AR, Willis KD, Braun SE, Rodin G, Lanoye A, Davies AE, Svikis D, Mazzeo S, Malkin M, Thacker L. Managing cancer and living meaningfully (CALM) in adults with malignant glioma: a proof-of-concept phase IIa trial. J Neurooncol. 2022 May;157(3):447-456. doi: 10.1007/s11060-022-03988-8. Epub 2022 Apr 18. PMID 35437687

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Therapy
Started | 14
Completed | 9
Not Completed | 5
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Therapy
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Recruitment for CALM
Description: Number of potential participants consented and enrolled
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Therapy
Number analyzed (Participants) | 14
Participants
  Consented | 14
  Enrolled | 14
  Started intervention | 12

2. Primary Outcome: Completion of CALM Sessions
Description: Number of participants completing CALM sessions
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Therapy
Number analyzed (Participants) | 12
Participants | 9

3. Primary Outcome: Post-session Assessment Completion
Description: Number of participants completing post-session surveys
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Therapy
Number analyzed (Participants) | 12
Participants | 10

4. Primary Outcome: Follow-up Assessment Completion
Description: Number of participants that completed a follow-up survey
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Therapy
Number analyzed (Participants) | 12
Participants | 4

5. Primary Outcome: Satisfaction With CALM Sessions
Description: Average rating of CALM session satisfaction score (average score across all participants following each CALM session multiple timepoints). Rating option is a range from 1 to 5 with 1 being not at all satisfied and 5 being very much satisfied. Higher scores indicate greater satisfaction.
Time Frame: Following each CALM session, every 2 weeks for 6 sessions: Weeks 2, 4, 6, 8, 10, and 12
Population: Of the 12 intervention initiators
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Therapy
Number analyzed (Participants) | 12
units on a scale | 4.6 [3 to 5]

6. Primary Outcome: Helpfulness of CALM Sessions
Description: Average rating of CALM session helpfulness score (average score across all participants following each CALM session multiple timepoints). Rating option is a range from 1 to 5 with 1 being not at all helpful and 5 being very much helpful. Higher scores indicate greater helpfulness.
Time Frame: Following each CALM session, every 2 weeks for 6 sessions: Weeks 2, 4, 6, 8, 10, and 12
Population: Of the 12 intervention initiators
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Therapy
Number analyzed (Participants) | 12
score on a scale | 4.6 [3 to 5]

7. Primary Outcome: Relevance of CALM
Description: Average rating of CALM session relevance score (average score across all participants following each CALM session multiple timepoints). Rating option is a range from 1 to 5 with 1 being not at all relevant and 5 being very much relevant. Higher scores indicate greater helpfulness.
Time Frame: Following each CALM session, every 2 weeks for 6 sessions: Weeks 2, 4, 6, 8, 10, and 12
Population: Of the 12 trial initiators
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Therapy
Number analyzed (Participants) | 12
score on a scale | 4.6 [2 to 5]

8. Primary Outcome: Utility of CALM
Description: Average rating of CALM session utility score (average score across all participants following each CALM session multiple timepoints). Rating option is a range from 1 to 5 with 1 being not at all useful and 5 being very much useful. Higher scores indicate greater helpfulness.
Time Frame: Following each CALM session, every 2 weeks for 6 sessions: Weeks 2, 4, 6, 8, 10, and 12
Population: of the 12 trial initiators
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Therapy
Number analyzed (Participants) | 12
score on a scale | 4.5 [3 to 5]

9. Primary Outcome: Intervention Satisfaction
Description: Mean rating of intervention satisfaction score (average score across all participants who completed the CALM intervention - one timepoint). Rating option is a range from 1 to 5 with 1 being not at all satisfied and 5 being very much satisfied. Higher scores indicate greater satisfaction.
Time Frame: 3 month - one timepoint
Population: of the 9 intervention completers
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Therapy
Number analyzed (Participants) | 9
score on a scale | 4.5 [3 to 5]

10. Primary Outcome: Number of Participants Likely to Recommend the Program to Others
Description: Rating of the likelihood of recommending the program to others.
Time Frame: 3 month timepoint
Population: of the 9 intervention completers
Measure: Count of Participants; unit: Participants
Arm/Group | Therapy
Number analyzed (Participants) | 9
Participants
  Will Recommend | 9
  Will not Recommend | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events and Serious adverse events were not collected for this trial.
Arm/Group | Therapy
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT04646213/Prot_SAP_001.pdf
  • Informed Consent Form (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT04646213/ICF_000.pdf